CLINICAL TRIAL: NCT04991116
Title: An Open-Label Extension Study to Evaluate Long Term Safety and Efficacy of Tildrakizumab in Patients With Psoriatic Arthritis.
Brief Title: Long Term Evaluation of Safety and Efficacy of Tildrakizumab in Patients With Psoriatic Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILD-21-01
Record Dates: First submitted 2021-07-29; First posted 2021-08-05 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TILD q12 weeks (Experimental)
  Interventions: Drug: TILD sub-cutaneous (SC) injection

INTERVENTIONS:
Drug: TILD sub-cutaneous (SC) injection — 1 mL injection of study medication

SUMMARY:
An open label phase 3 study

DETAILED DESCRIPTION:
Subjects from both INSPIRE 1 (TILD-19-07) and INSPIRE 2 (TILD-19-19) studies to roll over into this INSPIRE LTE study (TILD-21-01).

ELIGIBILITY:
Inclusion Criteria:

* Subjects possess the ability to understand the requirements of the study.
* Subject has provided written informed consent as evidenced by signature on an informed consent form approved by an institutional review board/EC.
* Agree to abide by the study restrictions, scheduled treatment, laboratory assessments, other study procedures and return to the site for the required assessments.
* Subject with PsA who had met all eligibility criteria for the parent study, had completed the parent study treatment period and has not developed any parent protocol criteria for premature discontinuation of treatment or withdrawal from the study.

Exclusion Criteria:

* Female subjects of childbearing potential who do not agree to abstain from heterosexual activity or practice a dual method of contraception.
* Female is pregnant or breastfeeding, or planning to become pregnant or initiate breastfeeding while enrolled in the study or up to 17 weeks after the last dose of IMP.
* Subject has previously been enrolled in this long-term extension study.
* Any condition that in the opinion of the Investigator represents an obstacle for study conduct and/or represents a potential unacceptable risk for the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and intensity of Adverse Events (AEs) recorded through the study period | Week 124
Proportion of Subject Who Reached (American College of Rheumatology Score of 20) ACR20 | Week 124
  ACR20 response is an aggregate of:
  1. at least 20% reduction in tender joint count and swollen joint count and at least 3 of the following 5 assessments:
  1. physician's global assessment of disease activity
  2. patient's global assessment of disease activity
  3. patient's assessment of pain
  4. patient's self-assessed disability based on health assessment questionnaire
  5. c-reactive protein
Proportion of Subjects Who Reached (American College of Rheumatology Score of 50) ACR50 | Week 124
  ACR50 response is an aggregate of:
  1. at least 50% reduction in tender joint count and swollen joint count and at least 3 of the following 5 assessments:
  1. physician's global assessment of disease activity
  2. patient's global assessment of disease activity
  3. patient's assessment of pain
  4. patient's self-assessed disability based on health assessment questionnaire
  5. c-reactive protein
Proportion of Subjects Who Reached (American College of Rheumatology Score of 70) ACR70 | Week 124
  ACR70 response is an aggregate of:
  1. at least 70% reduction in tender joint count and swollen joint count and at least 3 of the following 5 assessments:
  1. physician's global assessment of disease activity
  2. patient's global assessment of disease activity
  3. patient's assessment of pain
  4. patient's self-assessed disability based on health assessment questionnaire
  5. c-reactive protein

CONTACTS AND LOCATIONS:
Locations (103):
- United States (41):
  - Sunpharma site no 50, Dothan, Alabama
  - Sunpharma site no 80, Gilbert, Arizona
  - Sunpharma site no 65, Mesa, Arizona
  - Sunpharma site no 105, Phoenix, Arizona
  - Sunpharma site no. 30, Covina, California
  - Sunpharma site no 110, Encino, California
  - Sunpharma site no. 17, Fountain Valley, California
  - Sunpharma site no. 15, Thousand Oaks, California
  - Sunpharma site no 113, Avon Park, Florida
  - Sunpharma site no. 21, Clearwater, Florida
  - Sunpharma site no. 02, Hialeah, Florida
  - Sunpharma site no 71, Kissimmee, Florida
  - Sunpharma site no 107, Margate, Florida
  - Sunpharma site no. 05, New Port Richey, Florida
  - Sunpharma site no 32, Ocoee, Florida
  - SunPharma Site no 22, Tamarac, Florida
  - Sunpharma site no 52, Gainesville, Georgia
  - Sunpharma site no 51, Orland Park, Illinois
  - Sunpharma site no 49, Schaumburg, Illinois
  - Sunpharma site no 47, Skokie, Illinois
  - Sunpharma site no. 20, Wichita, Kansas
  - Sunpharma site no. 14, Springfield, Missouri
  - Sunpharma site no 104, St Louis, Missouri
  - Sunpharma site no 48, Kalispell, Montana
  - Sunpharma Site no 27, Lincoln, Nebraska
  - Sunpharma site no 33, Voorhees Township, New Jersey
  - Sunpharma site no 34, Charlotte, North Carolina
  - Sunpharma site no 111, Leland, North Carolina
  - Sunpharma site no 53, Wilmington, North Carolina
  - Sunpharma site no 35, Minot, North Dakota
  - Sunpharma site no. 11, Middleburg Heights, Ohio
  - Sunpharma site no 31, Greenville, South Carolina
  - Sunpharma site no. 08, Baytown, Texas
  - Sunpharma site no. 13, Baytown, Texas
  - Sunpharma Site no 28, Lubbock, Texas
  - Sunpharma site no 109, Mesquite, Texas
  - Sunpharma site no. 03, San Antonio, Texas
  - Sunpharma site no. 16, San Antonio, Texas
  - Sunpharma site no. 01, Tomball, Texas
  - Sunpharma site no 96, Salt Lake City, Utah
  - Sunpharma site no 66, Spokane, Washington
- Australia (3):
  - Sunpharma site no 59, Phillip, Australian Capital Territory
  - Sunpharma site no 58, Maroochydore, Queensland
  - Sunpharma site no. 24, Hobart, Tasmania
- Sunpharma site no 95, Trois-Rivières, Canada
- Czechia (4):
  - Sunpharma site no 36, Brno
  - Sunpharma site no 67, Prague
  - Sunpharma site no 89, Prague
  - Sunpharma site no 82, Zlín
- Estonia (3):
  - Sunpharma site no 44, Tallinn
  - Sunpharma site no 39, Tartu
  - Sunpharma site no 40, Tartu
- Germany (2):
  - Sunpharma site no 37, Berlin
  - Sunpharma site no 83, Herne
- India (10):
  - Sunpharma site no 92, Surat, Gujarat
  - Sunpharma site no 101, Belagavi, Karnataka
  - Sunpharma site no 91, Hubli, Karnataka
  - Sunpharma site no 108, Pune, Maharashtra
  - Sunpharma site no 100, Bangalore, Tamil Nadu
  - Sunpharma site no 93, Chennai, Tamil Nadu
  - Sunpharma site no 103, Chennai, Tamil Nadu
  - Sunpharma site no 114, Pune
  - Sunpharma site no 102, Secunderabad
  - Sunpharma site no 94, Sevilla
- Sunpharma site no 90, Verona, Italy
- Japan (10):
  - Sunpharma site no 73, Shinjuku-ku, Tokyo
  - Sunpharma site no 45, Fukuoka
  - Sunpharma site no 84, Itabashi-ku
  - Sunpharma site no 46, Kumamoto
  - Sunpharma site no 72, Mitaka
  - Sunpharma site no 79, Miyazaki
  - Sunpharma site no 78, Nagoya
  - Sunpharma site no 64, Sendai
  - Sunpharma site no 63, Sendai
  - Sunpharma site no 87, Tsu
- Poland (11):
  - Sunpharma site no 43, Bialystok
  - Sunpharma site no 69, Bialystok
  - Sunpharma site no 56, Krakow
  - Sunpharma site no 81, Lublin
  - Sunpharma site no 55, Nadarzyn
  - Sunpharma site no 106, Olsztyn
  - Sunpharma site no 85, Poznan
  - Sunpharma site no 68, Poznan
  - Sunpharma site no 60, Torun
  - Sunpharma site no 61, Warsaw
  - Sunpharma site no 112, Wroclaw
- Slovakia (3):
  - Sunpharma site no 74, Martin
  - Sunpharma site no 42, Nové Mesto nad Váhom
  - Sunpharma site no 41, Rimavská Sobota
- South Korea (2):
  - Sunpharma site no 98, Seoul
  - Sunpharma site no 70, Seoul
- Spain (7):
  - Sunpharma site no 57, A Coruña
  - SunPharma Site No 23, Córdoba
  - Sunpharma site no 38, Córdoba
  - Sunpharma site no 86, Málaga
  - Sunpharma site no 88, Santiago de Compostela
  - Sunpharma site no 62, Seville
  - Sunpharma site no 97, Valencia
- Taiwan (5):
  - Sunpharma site no 76, Kaohsiung City
  - Sunpharma site no 54, Taichung
  - Sunpharma site no 99, Taichung
  - Sunpharma site no 75, Tainan
  - Sunpharma site no 77, Taipei

IPD SHARING:
Plan to Share IPD: No